CLINICAL TRIAL: NCT01103024
Title: A 34-week Extension to a 28-week Multicenter, Randomized, Double-masked, Placebo Controlled, Dose-ranging Phase III Study to Assess AIN457 Versus Placebo in Inducing and Maintaining Uveitis Suppression in Adults With Active, Non-infectious, Intermediate, Posterior, or Panuveitis Requiring Immunosuppression (INSURE Study)
Brief Title: Extension Study to Assess Safety and Efficacy of AIN457 in Patients With Active Non-infectious Uveitis
Acronym: INSURE
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Core study in non-infectious active uveitis was terminated
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAIN457C2302E1; 2009-015509-38 (EudraCT Number)
Record Dates: First submitted 2010-04-09; First posted 2010-04-13 (Estimated); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Uveitis
Keywords: Active uveitis; intermediate uveitis; panuveitis; posterior uveitis; uveitis
MeSH Terms: conditions — Uveitis; Uveitis, Intermediate; Panuveitis; Uveitis, Posterior | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AIN457 300mg s.c every 2 weeks (Experimental)
  Interventions: Biological: AIN457
- AIN457 300mg s.c every 4 weeks (Experimental)
  Interventions: Biological: AIN457
- AIN457 150mg s.c every 4 weeks (Experimental)
  Interventions: Biological: AIN457
- Placebo s.c every 2 weeks (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: AIN457
  Arms: AIN457 300mg s.c every 2 weeks
Biological: AIN457
  Arms: AIN457 300mg s.c every 4 weeks
Biological: AIN457
  Arms: AIN457 150mg s.c every 4 weeks
Biological: Placebo
  Arms: Placebo s.c every 2 weeks

SUMMARY:
The purpose of the extension study was to provide patients completing the 28-week core study (NCT01095250) with an opportunity to receive an additional 22 weeks of continuous treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed the entire treatment period of the 28-week core study
* Patients must be able to understand and communicate with the investigator and comply with the requirements for the study and must give a written, signed, and dated informed consent before study treatment in the extension study

Exclusion Criteria:

* Inability or unwillingness to undergo repeated subcutaneous injections
* Inability to comply with study or follow-up procedures
* Any medical or psychiatric condition which, in the investigator's opinion would preclude the participant from adhering to the protocol or completing the study per protocol
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/mL)
* Women of childbearing potential (WoCBP), defined as all women physiologically capable of becoming pregnant, UNLESS
* They are using simultaneously double barrier or two acceptable methods of contraception
* They are postmenopausal with an appropriate clinical profile and had no regular menstrual bleeding for at least twelve (12) months prior to initial dosing
* They have undergone reliable surgical sterilization at least six (6) months prior to initial dosing
* Their career, lifestyle, or sexual orientation precludes intercourse with a male partner
* Partners have been sterilized by vasectomy or other reliable means

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-12; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Rate of recurrence | baseline to 52 weeks

SECONDARY OUTCOMES:
Change in immunosuppressive medication score from core study baseline | baseline to 52 weeks
Time to recurrence after the initial induction of quiescence (≤ 0.5+ anterior chamber cell grade and ≤ 0.5+ vitreous haze grade) by study treatment or rescue medication | baseline to 52 weeks
Mean change in best corrected visual acuity from baseline | baseline to 52 weeks
Change from baseline in Quality of Life/Patient reported outcome assessments | baseline to 52 weeks
Mean change in vitreous haze grade and anterior chamber cell grade from baseline to 52 weeks | baseline to 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- Texas Retina Associates, Arlington, Texas, United States
- Canada (2):
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, North York, Ontario
- Novartis Investigative Site, Ramat Gan, Israel
- Japan (6):
  - Novartis Investigative Site, Bunkyō City
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Fukushima
  - Novartis Investigational Site, Kyoto
  - Novartis Investigative Site, Sapporo
  - Novartis Investigative Site, Tochigi
- Novartis Investigative Site, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com